CLINICAL TRIAL: NCT03985241
Title: Functional Assessment of Myocardial Ischemia by Intracoronary Electrocardiogram
Acronym: FFRicECG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016-00726
Record Dates: First submitted 2019-06-05; First posted 2019-06-13 (Actual); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Coronary Artery Disease; Stable Angina; Coronary Artery Stenosis; Ischemia
Keywords: Intracoronary Electrocardiogram; Fractional Flow Reserve; Collateral Flow Index; Dobutamine
MeSH Terms: conditions — Coronary Artery Disease; Angina, Stable; Coronary Stenosis; Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Functional Assessment of Myocardial Ischemia by icECG (Experimental): Evaluation of ST-Shifts in the icECG acquired downstream of a coronary lesion during pharmacologic inotropic stress using dobutamine (40mcg/kg/min).
  Interventions: Diagnostic Test: Functional Assessment of Myocardial Ischemia by icECG

INTERVENTIONS:
Diagnostic Test: Functional Assessment of Myocardial Ischemia by icECG

SUMMARY:
In patients with chronic stable coronary artery disease (CAD), percutaneous coronary intervention (PCI) targets hemodynamically significant coronary lesions, i.e., those thought to cause inducible ischemia. The hemodynamic severity of a coronary stenosis increases with its tightness and with the myocardial mass of viable myocardium downstream of the stenosis.

Compared to the traditional anatomic angiographic approach, assessment of functional relevance by fractional flow reserve (FFR) during coronary angiography has been suggested to improve patient outcomes. Fractional flow reserve (FFR) is based on determination of the coronary perfusion pressure downstream of a stenosis during pharmacologic hyperemia. However, FFR relies on oversimplified physiologic concepts, which limits its usefulness in defining a true ischemic threshold. Furthermore, visual angiographic assessment continues to dominate the treatment decisions for intermediate coronary lesions.

Conversely, the intracoronary ECG (icECG) provides an inexpensive, sensitive and direct measure of myocardial ischemia. The icECG is easily acquired by attaching a reusable alligator clamp to a conventional angioplasty guidewire (at one tenth the price of a pressure sensor guidewire). The coronary guide wire positioned downstream of a coronary stenosis then acts as the exploring electrode. During pharmacologic stress, the icECG can provide direct evidence for regional myocardial ischemia to define the ischemic threshold in different types of coronary artery disease.

DETAILED DESCRIPTION:
INVASIVE PRESSURE-DERIVED INDICES OF STENOSIS SEVERITY

In the setting of stable coronary artery disease (CAD), PCI or coronary artery bypass grafting (CABG) targets coronary lesions causing inducible myocardial ischemia. With the advancement of technology, the development of a coronary pressure guide wire enabled to reliably measure coronary perfusion pressure downstream of a stenosis and therefore trans-stenotic pressure gradients. On the basis of comparisons to noninvasive stress tests, the concept of fractional flow reserve (FFR) was introduced. FFR determines the ratio of mean distal coronary pressure and mean aortic pressure (the effective coronary perfusion pressure) during (pharmacologic) hyperemia. A FFR value of near 1 is then equivalent to a totally normal coronary artery, whereas a cutoff of 0.75-0.80 is commonly used to determine that PCI is warranted.

With FFR, pharmacologic hyperemia is mandatory to induce minimal and constant myocardial resistance, which is the basis to directly relate coronary pressure and flow.In contrast, the recently introduced concept of the instantaneous wave-free ratio (iFR) claims to obviate the need for administration of pharmacologic stress. Instead, coronary pressure is analyzed at rest and during part of coronary diastole, when myocardial resistance is thought to be naturally constant and minimal (the so called wave-free period).

LIMITATIONS OF PRESSURE-DERIVED INDICES OF STENOSIS SEVERITY IN DEFINING THE ISCHEMIC THRESHOLD

A major limitation of pressure-derived indices of stenosis severity is related to the assumption of oversimplified physiologic concepts. Clinically, the diagnostic accuracy of FFR is restricted in three scenarios. Firstly, the pressure gradient evaluated by FFR is critically dependent on the magnitude of resistance offered by the microcirculation. With microvascular dysfunction, microvascular resistance remains inadequately high during pharmacologic hyperemia, meaning that the pressure gradient across the stenosis does not reflect the epicardial stenosis severity (overestimation of FFR).

Secondly, with a focal stenosis, but well-preserved microvascular function and minimal diffuse atherosclerosis, hyperemic coronary flow (although reduced) may still be above the ischemic threshold, although the pressure gradient suggests otherwise. Thirdly, with severe diffuse coronary atherosclerosis, coronary flow may be reduced below the ischemic threshold, but with only an insignificant fall in the hyperemic pressure gradient (FFR). In summary, although FFR claims otherwise, the ischemic threshold set by FFR is unreliable in a significant proportion of pathophysiological and clinical scenarios.

DIRECT ASSESSMENT OF REVERSIBLE MYOCARDIAL ISCHEMIA BY INTRACORONARY ELECTROCARDIOGRAM

The electrocardiogram (ECG) is an indispensable tool in the diagnosis of myocardial ischemia. The commonly used surface ECG is however limited especially in detecting short-lasting, or minor myocardial ischemia. Furthermore, ischemia in the territory of the left circumflex coronary artery is often undetected. Conversely, due to its close vicinity to the myocardium, the intracoronary ECG (icECG) is much more sensitive in detecting acute myocardial ischemia. The icECG is obtained by attaching a reusable alligator clamp to a coronary guidewire. With the guidewire positioned in a coronary artery, the derived (pseudo)unipolar icECG reflects local epicardial ECG.

The value of the icECG was first shown by Friedman et al. Unipolar icECG was recorded during balloon dilatation of coronary stenosis from the guidewire positioned across the stenosis to be dilated. Ischemic changes in icECG was observed in 72% of stenoses dilated. In the cases with no ischemic changes, either a prior myocardial infarction in the territory undergoing balloon dilatation or angiographic collaterals were present, consistent with the notion that ischemia was not inducible in nonviable myocardium or prevented by sufficient collaterals. Of note, ST changes in the surface ECG were seen in only 31% of cases.

With acute and complete coronary occlusion, perfusion to the dependent territory is usually severely reduced which explains the frequent occurrence of icECG changes. However, the usefulness of the icECG has also been shown with partial coronary occlusion. Experimentally, Battler et al. demonstrated that during a partial stenosis producing only mild regional dysfunction, significant ST segment changes in regional epicardial ECG could be observed after 2-3 minutes. Clinically, Hishikari et al. showed in patients with non-ST-segment elevation myocardial infarction (NSTEMI) that ST-segment-elevation in the icECG (icECG-STE) was observed in 27.6% of patients before PCI and was more common with LCX culprit lesions. Furthermore, in multivariate analysis, icECG-STE predicted greater peak values of troponin levels, consistent with greater myocardial injury. Similarly, but in patients undergoing elective PCI, Uetani et al. showed that icECG provided a useful method to predict post-procedural myocardial injury.

With regard to detection of inducible ischemia by pharmacologic (vasodilator) stress, Balian et al. compared STsegment shift in the icECG (IST) during intravenous adenosine infusion with FFR in 48 patients. 81% of patients with an FFR ≤0.80 showed IST during adenosine infusion, while 14% had IST with an FFR >0.80. As a major limitation, the study compared icECG findings only with FFR and therefore, the mechanism of discordant results remained unclear. Furthermore, the choice of the pharmacologic stressor was questionable: the perfusion abnormalities induced by adenosine are the result of flow heterogeneity, in contrast to exercise (or inotropic pharmacologic stress, eg. dobutamine), where the perfusion abnormalities are the result of myocardial ischemia (detectable by the electrocardiogram).

Thus, the goal of this study is to test the accuracy of intracoronary (ic) ECG during pharmacologic inotropic stress (i.e. Imitation of daily physical activity) to determine significant coronary lesions in comparison with established physiologic indices (fractional flow reserve (FFR), instantaneous wave-free ratio (iFR)) as well as with quantitatively determined percent diameter stenosis (%S) using biplane coronary angiography.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Referred for elective coronary angiography
* Written informed consent to participate in the study

Exclusion Criteria:

* Acute coronary syndrome
* Severe aortic stenosis
* Acute congestive heart failure NYHA III-IV
* Prior myocardial infarction in the vascular territory undergoing pressure measurements
* Presence of left bundle branch block, non-sinus rhythm or paced rhythm in resting ECG
* Coronary anatomy unsuitable for coronary pressure measurements
* Severe pulmonary, renal or hepatic disease
* Contraindication to inotropic stress
* Women of childbearing age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-12-03 (Actual); Primary Completion 2019-12-13 (Actual); Study Completion 2019-12-13 (Actual)

PRIMARY OUTCOMES:
Intracoronary Electrocardiogram ST-Segment Shift | Measured at maximal heart frequency (=~6min after begin dobutamine)
  Change in intracoronary ST-segment shift from baseline to hyperemia, measured at the J-Point in mV

SECONDARY OUTCOMES:
Percent Diameter Stenosis | During diagnostic angiography at the beginning of the coronary angiography
  Assessment of percent diameter Stenosis using quantitative coronary angiography; comparison with icECG
Fractional Flow Reserve | Measured at maximal heart frequency (=~6min after begin dobutamine)
  FFR during steady-state hyperemia; comparison with icECG
Instantaneous wave-free ratio | Measured at baseline before inotropic stress
  iFR at baseline; comparison with icECG
Area at Risk | Measured after the coronary angiography, expected to be on average after 3 days
  Myocardial area at risk in percent using the Approach-Score and relation to intracoronary ECG ST-Segment shift

CONTACTS AND LOCATIONS:
Overall Officials: Christian Seiler, MD, Prof, Principal Investigator — Inselspital, Bern University Hospital
Locations (1):
- University Hospital Inselspital, Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Friedman et al. Circulation 1986 - Value of the intracoronary electrocardiogram to monitor myocardial ischemia during percutaneous transluminal coronary angioplasty. — https://www.ncbi.nlm.nih.gov/pubmed/2942314
- See also: de Marchi et al. JACC 2012 - Determinants of prognostically relevant intracoronary electrocardiogram ST-segment shift during coronary balloon occlusion. — https://www.ncbi.nlm.nih.gov/pubmed/22835408